CLINICAL TRIAL: NCT01338103
Title: Treatment of Moderate to Severe Patients With Pemphigus With the Monoclonal Anti CD20 Antibody Rituximab at a Protocol of 1000mgX2 and Assessment of Their Immune Status Via the Cylex Test
Brief Title: Treatment of Pemphigus Patients With Rituximab 1000mgX2 and Assessment of Immune Status Via Cylex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Leumit Health Services (Other)
Responsible Party: Daniel Mimouni MD, Rabin Medical Center, Department of Dermatology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5474
Record Dates: First submitted 2011-04-17; First posted 2011-04-19 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-03

CONDITIONS: Pemphigus
Keywords: Pemphigus; Rituximab; Cylex
MeSH Terms: conditions — Pemphigus | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — intravenous (IV) Rituximab 1 gramX2, every (q) 2 weeks.

SUMMARY:
The purpose of this study is to determine whether Rituximab, in the same doses as used in rheumatoid arthritis patients, will benefit pemphigus patients. It also tests immune function via the Cylex assay in pemphigus patients before and after treatment with RItuximab.

ELIGIBILITY:
Inclusion Criteria:

1. Pemphigus patients with moderate-severe disease

Exclusion Criteria:

1. Pregnancy or lactation
2. Woman of reproductive age not using birth control measures.
3. Prior severe allergy or anaphylaxis with a human monoclonal antibody
4. Heart failure
5. Unstable angina or ischemic heart disease
6. Uncontrolled arrhythmia
7. HIV positive
8. Active hepatitis B infection or positive for hepatitis C virus (HCV) antibodies.
9. Severe dementia or a psychiatric illness
10. Active acute infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Complete or partial remission off treatment (based on the consensus statement for pemphigus) | 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Bullous diseases clinic, Department of dermatology, Rabin Medical Center, Petah Tikva, Israel